CLINICAL TRIAL: NCT06744894
Title: Selinexor Combined With Ixazomib and Lenalidomide as Maintenance Therapy in Patients With Multiple Myeloma
Brief Title: SIL as Maintenance Therapy in Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Associate Chief Physician, Associate Professor, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIL2024
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Maintenance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maintenance Therapy (Experimental): Patients were treated by Selinexor combined with Ixazomib and Lenalidomide as Maintenance Therapy
  Interventions: Drug: Selinexor combined with Ixazomib and Lenalidomide as Maintenance Therapy

INTERVENTIONS:
Drug: Selinexor combined with Ixazomib and Lenalidomide as Maintenance Therapy — Patients were treated by Selinexor (40mg po qw d1-28) combined with Ixazomib (4mg po on days 1, 8, and 15 in 28-day cycles) and Lenalidomide(10mg po qd d1-21) as Maintenance Therapy.

SUMMARY:
The goal of this phase 2 trial is to test the safety and efficacy of selinexor combined with ixazomib and lenalidomide as maintenance therapy in patients with multiple myeloma.

DETAILED DESCRIPTION:
The investigators will evaluate safety and efficacy of selinexor combined with ixazomib and lenalidomide as maintenance therapy in patients with multiple myeloma post complete remission. Event-free survival (EFS), progression-free survival (PFS), overall survival (OS), adverse events (AEs) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Multiple Myeloma according World Health Organization (WHO) classification;
* Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
* Patient must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted;
* Patient is willing and able to adhere to the study visit schedule and other protocol requirements;
* Documented response to ASCT (PR, VGPR, CR/stringent complete response [sCR]) according to IMWG criteria.

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment.
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy.
* Pregnant or lactating women

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  PFS was defined as the time from study entry until disease progression

SECONDARY OUTCOMES:
EFS | 2 years
  EFS was defined as the time from treatment initiation to progression, relapse, new treatment, or death by any cause, whichever occurred first.
OS | 2 years
  OS was defined as the time from treatment initiation to death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, PhD, Principal Investigator — Navy General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No